CLINICAL TRIAL: NCT06747325
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Fei Re Qing Granules in the Treatment of Elderly Community-Acquired Pneumonia
Brief Title: Clinical Trial of Fei Re Qing Granules in the Treatment of Elderly Community-Acquired Pneumonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: Third Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Henan university of CM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM for Elderly CAP
Record Dates: First submitted 2024-12-14; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Community-Acquired Pneumonia (CAP)
Keywords: elderly community-acquired pneumonia (CAP); traditional Chinese medicine; randomized controlled trial; Fei Re Qing Granules
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): The patients in the trial group received routine standard treatments, and oral Fei Re Qing Granules (One bag/time, 3 times/day).
  Interventions: Drug: Fei Re Qing Granules; Other: Routine standard treatments
- Control group (Placebo Comparator): The patients in the control group received routine standard treatments, and Placebo granules
  Interventions: Other: Routine standard treatments; Drug: Placebo granules

INTERVENTIONS:
Drug: Fei Re Qing Granules — Fei Re Qing Granules (Ingredients: Scutellaria baicalensis [Huang Qin], Trichosanthes kirilowii [Gua Lou], Forsythia suspensa [Lian Qiao], Fritillaria thunbergii [Zhe Bei Mu], etc.)
  Arms: Test group
Other: Routine standard treatments — Routine standard treatments
Drug: Placebo granules — The placebo granules are prepared using 5% of the active drug, ensuring consistency in appearance, weight, color, and odor with the Fei Re Qing Granules
  Arms: Control group

SUMMARY:
This study aims to evaluate the clinical efficacy of traditional Chinese medicine formula granules (Fei Re Qing Granules) in the treatment of elderly community-acquired pneumonia, establish a treatment protocol, and obtain high-level clinical evidence.

DETAILED DESCRIPTION:
This study evaluates the efficacy and safety of Fei Re Qing Granules for elderly community-acquired pneumonia (CAP) through a multicenter, randomized, double-blind, placebo-controlled trial.

Key elements of the trial include:

Design: Conducted across multiple centers, comparing treatment and placebo groups.

Participants: Patients aged 65-80 years diagnosed with CAP according to both Western and Traditional Chinese Medicine (TCM) diagnostic criteria.

Intervention:

Test group: Fei Re Qing Granules administered alongside standard CAP treatments.

Control group: Placebo granules matching the appearance and composition of the active granules, plus standard treatments.

Outcomes:

Primary efficacy indicator: Time to clinical stability. Secondary indicators: Symptom improvement, hospital stay length, and imaging-based inflammation resolution.

TCM-specific indicators assess syndrome improvements and integrate modern scoring methods (e.g., CURB-65).

Study Duration: Two 7-day treatment cycles with 12-week follow-ups. This trial seeks to establish robust evidence for integrating Fei Re Qing Granules into TCM-based CAP management strategies

ELIGIBILITY:
Inclusion Criteria:

* Inpatients diagnosed with community-acquired pneumonia (CAP) according to the diagnostic criteria.
* Diagnosed with Phlegm-Heat Obstructing the Lungs syndrome based on Traditional Chinese Medicine (TCM).
* Aged ≥65 and ≤80 years, regardless of gender.
* Onset of illness within 72 hours.
* Clinical symptoms must include at least two of the following four primary。symptoms: cough, sputum production, dyspnea, and pleuritic chest pain.
* Voluntary participation and signed informed consent.

Exclusion Criteria:

* Patients with altered mental status, consciousness disorders, dementia, or psychiatric disorders.
* Patients requiring invasive mechanical ventilation or endotracheal intubation.
* Patients with conditions such as pleural effusion, bronchiectasis, active pulmonary tuberculosis, pulmonary abscess, lung cancer, asthma, or chronic obstructive pulmonary disease (COPD).
* Patients with neuromuscular diseases or those bedridden for long periods, posing a risk of aspiration.
* Patients with cancer, severe cardiovascular diseases (acute myocardial infarction, heart failure stage III or above), or severe liver and kidney diseases (e.g., cirrhosis, portal hypertension with variceal bleeding, dialysis, or kidney transplantation).
* Patients participating in other drug clinical trials or known to be allergic to the study medication.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Stability | From the start of treatment, the time is recorded until the patient reaches clinical stability, whichever came first, assessed up to 2 weeks.
  The criteria for clinical stability require meeting all five of the following indicators:
  Body temperature ≤ 37.8°C for more than 24 hours; Resting heart rate ≤ 100 beats per minute; Resting respiratory rate ≤ 24 breaths per minute; Systolic blood pressure ≥ 90 mmHg; Oxygen saturation (SpO₂) ≥ 90% (or arterial oxygen partial pressure ≥ 60 mmHg on room air).
  During the treatment period, log cards will be issued to monitor and record vital signs (temperature, respiration, blood pressure, heart rate, and SpO₂) every 12 hours. The time to clinical stability will be calculated based on these records

SECONDARY OUTCOMES:
Improvement of Clinical Symptoms | Evaluations will be conducted on Day 0, Day 4, Day 7, Day 14 (or at discharge) and during follow-up at 4 weeks and 12 weeks.
  Improvement in clinical symptoms is defined as at least two of the four main clinical symptoms (cough, sputum production, pleuritic chest pain, and dyspnea) showing an improvement of at least one grade, with no worsening of the other symptoms.
  The grade of clinical symptoms is divided into four levels:
  None Mild Moderate Severe The number of cases with clinical symptom improvement is calculated as the ratio of improved cases to the total cases in each group.
Length of Hospital Stay | From the start of treatment, the time is recorded until the patient discharge, whichever came first, assessed up to 2 weeks.
  The length of hospital stay is calculated as the number of days from admission to when the patient meets the discharge criteria.
  Discharge Criteria include:
  Body temperature normal for more than 24 hours; Resting heart rate ≤ 100 beats/min; Resting respiratory rate ≤ 24 breaths/min; Systolic blood pressure ≥ 90 mmHg; Oxygen saturation ≥ 90% (or arterial oxygen partial pressure ≥ 60 mmHg on room air).
  If the patient can be transitioned to oral medication and does not require further management for complications or mental disorders, discharge may be considered.
Confusion, Urea, Respiratory rate, Blood pressure, and Age ≥65 Score (CURB-65 score). | The CURB-65 score is assessed on Day 0, Day 4, Day 7, Day 14 (or at discharge) and during follow-up at 4 weeks and 12 weeks.
  The Confusion, Urea, Respiratory rate, Blood pressure, and Age ≥65 Score (CURB-65 score) is a clinical tool used to assess the severity of community-acquired pneumonia (CAP) and the associated mortality risk based on five clinical indicators(On a 5-point scale, 5 is the worst and 0 is the best.):
  Confusion (assessed by changes in mental status) ：0-5 score Urea (blood urea nitrogen level >7 mmol/L) ：0-5 score Respiratory rate (≥30 breaths/min) ：0-5 score Blood pressure (systolic BP <90 mmHg or diastolic BP ≤60 mmHg) ：0-5 score Age (≥65 years) ：0-5 score The total score is calculated by adding points for each indicator, with a higher score indicating more severe disease and higher risk of mortality.
Traditional Chinese Medicine Syndrome Efficacy Evaluation | These evaluations will be carried out on Day 0, Day 4, Day 7, Day 14 (or at discharge).
  Based on the Guidelines for Clinical Research of Traditional Chinese Medicine New Drugs, each symptom is rated on a scale of None, Mild, Moderate, and Severe (4 levels).
  Primary symptoms (e.g., cough, sputum production, chest pain, and dyspnea) are scored 0, 2, 4, and 6 points, respectively.
  Secondary symptoms (e.g., fever, thirst, flushed face, yellow urine, constipation, and abdominal distention) are scored 0 or 1 point, depending on their presence or absence.
  For the Phlegm-Heat Obstructing the Lungs syndrome, the overall score is calculated by summing the points for primary and secondary symptoms before and after treatment. The treatment outcomes are classified into four levels:
  Clinical Recovery: Syndrome score reduction ≥95%. Significant Improvement: Syndrome score reduction ≥70%. Effective: Syndrome score reduction ≥30%. Ineffective: Syndrome score reduction <30%.
Comprehensive Clinical Efficacy Assessment | This evaluation will be conducted on Day 14 (or at discharge).
  Based on the Antimicrobial Drug Clinical Research Guidelines, the efficacy is classified into four levels:
  Clinical Recovery: At the end of treatment, the patient's clinical symptoms, signs, major laboratory tests, and microbiological tests have all returned to normal.
  Significant Improvement: At the end of treatment, the patient's condition has noticeably improved, but one of the four key indicators (symptoms, signs, laboratory tests, or microbiological tests) has not fully returned to normal.
  Progress: At the end of treatment, the patient's condition has shown some improvement, but not enough to be considered significant.
  Ineffective: At the end of treatment, the patient's condition has not improved or has worsened.
Modified Pneumonia Imaging Absorption Evaluation Scale | The evaluations will be conducted on Day 0, Day 7 (or at discharge), and at 12 weeks during follow-up.
  Chest imaging examinations will be performed on both groups of subjects before and after treatment, as well as at the end of the follow-up, to observe the changes in lung imaging. The degree of pneumonia absorption will be recorded using the evaluation scale.
  Evaluation Process: Two radiology experts will independently assess and score the imaging results, and the average score will be taken.
  Assessment Points: The evaluations will be conducted on Day 0, Day 7 (or at discharge), and at 12 weeks during follow-up.
  This method helps assess the extent of pneumonia absorption and track changes in lung conditions over time.
Pathogen Clearance Rate | This will be assessed at pre-treatment, Day 7, Day 14 (or at discharge) for each patient.
  The microbiological results of both groups of patients during hospitalization will be recorded. Pathogen clearance is defined as follows:
  Clearance: If no pathogen is detected in more than three consecutive tests. Replacement: If the original pathogen is no longer detected and a new pathogen is identified.
  Not cleared: If the pathogen load does not decrease, or although the pathogen load has decreased, it has not been completely cleared.
Readmission Rate | The readmission rate will be assessed at 4 weeks and 12 weeks during follow-up, with a detailed record of the reasons for readmission.
  The readmission rate includes the all-cause readmission rate and pneumonia-related readmission rate:
  All-cause readmission refers to patients being readmitted for any disease, with the admission criteria based on relevant disease guidelines.
  Pneumonia-related readmission refers to patients being readmitted due to a recurrent lung infection, with admission criteria based on the "Chinese Guidelines for the Diagnosis and Treatment of Adult Community-Acquired Pneumonia (2016 edition)", using the CURB-65 score to determine the need for hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, Doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine